CLINICAL TRIAL: NCT03027245
Title: Incidence and Resolution of Eribulin-Induced Peripheral Neuropathy (IRENE)
Brief Title: Incidence and Resolution of Eribulin-Induced Peripheral Neuropathy
Acronym: IRENE
Status: Completed | Type: Observational
Sponsor: Eisai GmbH (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Other Study IDs: E7389-M044-504
Record Dates: First submitted 2017-01-19; First posted 2017-01-23 (Estimated); Last update posted 2022-07-13 (Actual); Status verified 2022-03

CONDITIONS: Locally Advanced or Metastatic Breast Cancer
Keywords: locally advanced or metastatic breast cancer; peripheral neuropathy; chemotherapy-induced peripheral neuropathy; eribulin
MeSH Terms: conditions — Breast Neoplasms; Peripheral Nervous System Diseases | interventions — eribulin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Eribulin-treated participants: Participants treated with eribulin according to Fachinformation and managed according to clinical practice
  Interventions: Drug: Eribulin

INTERVENTIONS:
Drug: Eribulin

SUMMARY:
Study E7389-M044-504 is an observational, post-authorization, single-arm, prospective, multicenter cohort study conducted to characterize and determine the incidence of eribulin-induced peripheral neuropathy (PN), and the frequency and time to resolution of eribulin-induced PN in adult participants treated with eribulin in a real-life setting with locally advanced or metastatic breast cancer (MBC) who have progressed following at least one and up to three chemotherapeutic regimens for advanced disease.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced or MBC with progression after at least one chemotherapeutic regimen for advanced disease eligible for treatment with eribulin according to Fachinformation. Prior therapy should have included an anthracycline and a taxane in either the adjuvant or metastatic setting unless participants were not suitable for these treatments
* 1-3 prior chemotherapeutic regimens for advanced disease
* Age >=18 years at the time of Informed Consent
* Ability to understand and willingness to respond to questions related to their health
* Decision for the participant to start treatment with eribulin has been made prior to inclusion in this study.
* Signed written Informed Consent

Exclusion Criteria:

* Previous treatment with eribulin in any line of treatment
* Contraindication according to the Fachinformation of eribulin
* Pregnancy or lactation
* Participation in an interventional clinical trial at the same time

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female participants greater than or equal to (>=) 18 years with locally advanced or MBC
Sampling Method: Probability Sample
Enrollment: 353 (Actual)
Dates: Start 2016-10-13 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Number of participants experiencing eribulin-induced peripheral neuropathy (PN) | Approximately 15 months, or until death or resolution of peripheral neuropathy, or return to baseline level, whichever comes first
Percentage of participants experiencing eribulin-induced PN | Approximately 15 months, or until death or resolution of peripheral neuropathy, or return to baseline level, whichever comes first
Number of participants with the indicated grade of eribulin-induced PN, as determined by Common Terminology Criteria for Adverse Events (CTCAE), grade version 4.0 | Approximately 15 months, or until death or resolution of peripheral neuropathy, or return to baseline level, whichever comes first
Percentage of participants who experienced dose modifications of eribulin treatment due to eribulin-induced PN | Approximately 15 months, or until death or resolution of peripheral neuropathy, or return to baseline level, whichever comes first
Percentage of participants who discontinued eribulin treatment due to eribulin-induced PN | Approximately 15 months, or until death or resolution of peripheral neuropathy, or return to baseline level, whichever comes first
Time to eribulin treatment discontinuation due to eribulin-induced PN | Approximately 15 months, or until death or resolution of peripheral neuropathy, or return to baseline level, whichever comes first
Number of resolved cases in participants who experience eribulin-induced PN | Approximately 15 months, or until death or resolution of peripheral neuropathy, or return to baseline level, whichever comes first
  A resolved case is defined as one that ended or returned to baseline as determined by CTCAE grade version 4.0
Percentage of resolved cases in participants who experience eribulin-induced PN | Approximately 15 months, or until death or resolution of peripheral neuropathy, or return to baseline level, whichever comes first
  A resolved case is defined as one that ended or returned to baseline as determined by CTCAE grade version 4.0
Time to resolution of eribulin-induced PN | Approximately 15 months, or until death or resolution of peripheral neuropathy, or return to baseline level, whichever comes first
  Time to resolution is defined as the time from onset (or worsening from baseline) to the date of resolution (defined as stop of PN or return to baseline), as determined by CTCAE grade version 4.0.
Number of therapeutic interventions (e.g., analgesics) being used to treat eribulin-induced PN | Approximately 15 months, or until death or resolution of peripheral neuropathy, or return to baseline level, whichever comes first

SECONDARY OUTCOMES:
Health-related quality of life scores measured using the Patient Neurotoxicity Questionnaire | Approximately 15 months, or until death or resolution of peripheral neuropathy, or return to baseline level, whichever comes first
Health-related quality of life scores measured using the EuroQOl-5 Dimensions-3 Levels (EQ-5D-3L) questionnaire | Approximately 15 months, or until death or resolution of peripheral neuropathy, or return to baseline level, whichever comes first
Time to disease progression | Approximately 15 months, or until death or resolution of peripheral neuropathy, or return to baseline level, whichever comes first
  Time to disease progression is defined as the time from the start of eribulin treatment to Investigator assessment of disease progression (clinical or radiological)
Number of participants with any serious adverse event (SAE) and number of participants with any non-serious AE | Approximately 15 months, or until death or resolution of peripheral neuropathy, or return to baseline level, whichever comes first
Percentage of participants with any SAE and percentage of participants with any non-serious AE | Approximately 15 months, or until death or resolution of peripheral neuropathy, or return to baseline level, whichever comes first

CONTACTS AND LOCATIONS:
Locations (65):
- Germany (65):
  - Eisai Trial Site 1, Amberg
  - Eisai Trial Site 1, Aschaffenburg
  - Eisai Trial Site 2, Aschaffenburg
  - Eisai Trial Site 1, Augsburg
  - Eisai Trial Site 2, Augsburg
  - Eisai Trial Site 1, Aurich
  - Eisai Trial Site 1, Berlin
  - Eisai Trial Site 2, Berlin
  - Eisai Trial Site 3, Berlin
  - Eisai Trial Site 1, Bonn
  - Eisai Trial Site 2, Bonn
  - Eisai Trial Site 1, Cologne
  - Eisai Trial Site 2, Cologne
  - Eisai Trial Site 1, Darmstadt
  - Eisai Trial Site 1, Donauwörth
  - EISAI Trial Site 1, Dresden
  - Eisai Trial Site 1, Düren
  - Eisai Trial Site 1, Essen
  - Eisai Trial Site 1, Esslingen am Neckar
  - Eisai Trial Site 1, Eutin
  - Eisai Trial Site 1, Freiburg im Breisgau
  - Eisai Trial Site 1, Fürstenwalde
  - Eisai Trial Site 1, Gelsenkirchen
  - Eisai Trial Site 1, Georgsmarienhütte
  - Eisai Trial Site 1, Greifswald
  - Eisai Trial Site 1, Hanover
  - Eisai Trial Site 2, Hanover
  - Eisai Trial Site 1, Hof
  - Eisai Trial Site 1, Homburg
  - Eisai Trial Site 1, Ilsede
  - Eisai Trial Site 1, Karlsruhe
  - Eisai Trial Site 1, Kassel
  - Eisai Trial Site 1, Kiel
  - Eisai Trial Site 2, Kiel
  - Eisai Trial Site 1, Koblenz
  - Eisai Trial Site 1, Lahr
  - Eisai Trial Site 1, Landshut
  - Eisai Trial Site 1, Lemgo
  - Eisai Trial Site 1, Lübeck
  - Eisai Trial Site 1, Magdeburg
  - Eisai Trial Site 1, Mainz
  - Eisai Trial Site 1, Mannheim
  - Eisai Trial Site 1, Marktredwitz
  - Eisai Trial Site 1, München
  - Eisai Trial Site 2, München
  - Eisai Trial Site 3, München
  - Eisai Trial Site 1, Münster
  - Eisai Trial Site 1, Naunhof
  - Eisai Trial Site 1, Nuremberg
  - Eisai Trial Site 1, Oberhausen
  - Eisai Trial Site 1, Offenbach
  - Eisai Trial Site 1, Offenburg
  - Eisai Trial Site 1, Oldenburg
  - Eisai Trial Site 1, Potsdam
  - Eisai Trial Site 1, Püttlingen
  - Eisai Trial Site 1, Quedlinburg
  - Eisai Trial Site 1, Rodgau
  - Eisai Trial Site 1, Rotenburg (Wümme)
  - Eisai Trial Site 1, Saarlouis
  - Eisai Trial Site 1, Stolberg
  - Eisai Trial Site 1, Stuttgart
  - Eisai Trial Site 2, Stuttgart
  - Eisai Trial Site 1, Tübingen
  - Eisai Trial Site 1, Villingen-Schwenningen
  - Eisai Trial Site 1, Worms

IPD SHARING:
Plan to Share IPD: No